CLINICAL TRIAL: NCT06868992
Title: Study of the Link Between Metabolic Dysfunction-Associated Steatohepatitis (MASH) and Mitochondria-Associated Membranes (MAMs) Alteration in Patients Undergoing Bariatric Surgery - MAMBA
Brief Title: Study of the Link Between MASH ( Metabolic Dysfunction-Associated Steatohepatitis) and MAMs (Mitochondria-Associated Membranes ) Alteration in Patients Undergoing Bariatric Surgery - MAMBA
Acronym: MAMBA
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_1096; 2024-A02591-46 (Other: ID-RCB)
Record Dates: First submitted 2025-03-03; First posted 2025-03-11 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease; Metabolic Dysfunction-Associated Steatohepatitis; Sleeve Gastrectomy; Gastric Bypass Surgery
Keywords: MASH; MASLD; Mitochondria-Associated Membranes (MAMs); Bariatric Surgery; Hepatic Fibrosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Bariatric Surgery; Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biobank (blood, urine, faeces) Tissue biobank (adipose tissue, muscle) Tissue biobank (liver)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bariatric Surgery Group: Patients with MASLD undergoing bariatric surgery (sleeve gastrectomy or gastric bypass) with an indication for liver biopsy due to suspected MASH
  Interventions: Procedure: Bariatric surgery (Sleeve Gastrectomy or Gastric Bypass)

INTERVENTIONS:
Procedure: Bariatric surgery (Sleeve Gastrectomy or Gastric Bypass) — Patients undergoin bariatric surgery with simultaneous liver biopsy to analyze MAMs alterations in liver and PBMCs. Follow-up assessments at 6 and 12 months.

SUMMARY:
The main research hypothesis is that alterations in the communication between the endoplasmic reticulum (ER) and the mitochondria at contact sites called mitochondria-associated membranes (MAMs) occurs in different hepatic cell types of patients with Metabolic Dysfunction-Associated Steatotic Liver Disease (MALSD) and is involved in the progression towards MASH and could also influence the process of improvement of MASH.

This study aims to investigate the link between Metabolic Dysfunction-Associated Steatohepatitis (MASH) and Mitochondria-Associated Membranes (MAMs) in liver cells and peripheral blood mononuclear cells (PBMCs) in patients undergoing bariatric surgery. The primary objective is to analyze MAMs alterations in hepatocytes in MASH patients compared to non-MASH patients. Secondary objectives include evaluating the correlation between MAMs in PBMCs and liver cells and assessing MAMs changes post-bariatric surgery.

ELIGIBILITY:
* Inclusion Criteria * :

  * Female or male adult patients
  * Patient who has benefited from a pluridisciplinary evaluation (medical, surgical, psychiatric), with a favorable opinion for a sleeve gastrectomy or a gastric bypass.
  * Patient with an indication Indication for intraoperative liver biopsy due to suspected MASH
  * Patient who agrees to be included in the study and who signs the informed consent form,
  * Patient affiliated to a healthcare insurance plan.
* Exclusion Criteria * :

  * Patient presenting Hepatitis B as defined as presence of hepatitis B surface antigen (HBsAg).
  * Patient presenting previous or current infection with Hepatitis C
  * Autoimmune hepatitis as defined by anti-nuclear antibody (ANA) of 1:160 or greater and liver histology consistent with autoimmune hepatitis or previous response to immunosuppressive therapy.
  * Patient presenting Autoimmune cholestatic liver disorders as defined by elevation of alkaline phosphatase and anti-mitochondrial antibody of greater than 1:80 or liver histology consistent with primary biliary cirrhosis or elevation of alkaline phosphatase and liver histology consistent with sclerosing cholangitis.
  * Patient presenting Wilson disease as defined by ceruloplasmin below the limits of normal and liver histology consistent with Wilson disease.
  * Patient presenting Alpha-1-antitrypsin deficiency as defined by alpha-1-antitrypsin level less than normal and liver histology consistent with alpha-1-antitrypsin deficiency.
  * Patient presenting Hemochromatosis as defined by presence of 3+ or 4+ stainable iron on liver biopsy and homozygosity for C282Y or compound heterozygosity for C282Y/H63D.
  * Patient presenting Drug-induced liver disease as defined on the basis of typical exposure and history.
  * Patient presenting Bile duct obstruction as shown by imaging studies.
  * History of ingestion of medications known to produce steatosis, such as corticosteroids, high-dose estrogen, tamoxifen, methotrexate, amiodarone or tetracycline in the previous 6 months.
  * Evidence of cirrhosis or previously known cirrhosis based on the results from previous liver biopsy or history of portal hypertension presented by ascites, hepatic encephalopathy or varices
  * Consommation régulière et/ou excessive d'alcool (plus de 30g/j pour les hommes et plus de 15 g/j pour les femmes) sur une période de plus de 2 ans au cours des 10 dernières années.
  * History of known HIV infection
  * History of type 1 diabetes
  * Pregnant women or breastfeeding mothers*.
  * Minor patient
  * Patient deprived of liberty,
  * Patients under psychiatric care
  * Patients admitted to a health or social care establishment for purposes other than research
  * Mentally unbalanced patients, under supervision or guardianship,
  * Patients not affiliated to a social security scheme or benefiting from a similar scheme
  * Patient who does not understand French/ is unable to give consent,
  * Patient already included in a trial who may interfere with the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with MASLD and obesity for whom an indication for bariatric surgery AND the indication for a per-procedure liver biopsy during bariatric surgery is indicated because of the suspected presence of MASH
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
MAMs alterations in hepatocytes | Baseline (T0)
  Number of MAM contacts in liver cells at baseline (T0)

SECONDARY OUTCOMES:
MAMs alterations in non-parenchymal liver cells (T0) | Baseline (T0)
  Number of MAM contacts in non-parenchymal liver cells at baseline (T0)
MAMs alterations in PBMCs (T0, T6, T12 months) | Baseline (T0) , T6, T12 months
  Number of MAM contacts in PBMCs
Changes in hepatic markers of MASLD post-surgery | T0 to T6, T6 to T12, T0 toT12 (months)
  Changes in measurements, of Vibration Controlled Transient Elastographt (VCTE) after bariatric surgery (∆T0-T6months, ∆T6-T12months and ∆T0-T12months).
Changes in hepatic markers of MASLD post-surgery (2) | T0 to T6, T6 to T12, T0 toT12 (months)
  Controlled attenuation Parameter (CAP), after bariatric surgery (∆T0-T6months, ∆T6-T12months and ∆T0-T12months).
Correlation between MASH improvement and MAMs changes | T0-T12 months
  Correlation between MASH improvement and MAMs changes

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hospices Civils de Lyon - Hôpital Edouard Herriot, Lyon, France
  - Centre Hospitalier Lyon Sud, Endocrinologie, Diabète et nutrition, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No